CLINICAL TRIAL: NCT03152240
Title: Coronary Anatomy Study and Times Since the Onset of Acute MyocardiaI Infarction Symptoms in Women Until the Opening of the Artery (TAPAC Study)
Brief Title: Coronary Anatomy Study and Times Since the Onset of Acute Myocardial Infarction Symptoms in Women Until the Opening of the Artery (TAPAC Study)
Acronym: TAPAC
Status: Completed | Type: Observational
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: TAPAC study
Record Dates: First submitted 2017-05-04; First posted 2017-05-12 (Actual); Last update posted 2019-02-27 (Actual); Status verified 2019-02

CONDITIONS: Myocardial Infarction
Keywords: Acute Coronary Syndrome; Primary Angioplasty; Gender
MeSH Terms: conditions — Myocardial Infarction; Acute Coronary Syndrome; Coitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Women patients: Women patients
  Interventions: Other: Non intervention
- Men patients: Men patients
  Interventions: Other: Non intervention

INTERVENTIONS:
Other: Non intervention — Non intervention

SUMMARY:
TAPAC study is an an investigator-driven, observational, prospective,cohort aimed at evaluating differences between men and women in patients undergoing primary angioplasty : hospital medical care, successful markers myocardial reperfusion and the anatomical substrate by describing the underlying coronary anatomy will be compared.

DETAILED DESCRIPTION:
TAPAC study is an an investigator-driven, observational, prospective,cohort aimed at evaluating differences between men and women in patients undergoing primary angioplasty : hospital medical care, successful markers myocardial reperfusion and the anatomical substrate by describing the underlying coronary anatomy will be compared.

ELIGIBILITY:
Inclusion Criteria:

Patients with:

* Aged 18 years or over.
* AMI (Acute Mycardial Infarction ) with ST segment elevation and indication of primary angioplasty in whom at least one diagnostic procedure with coronary angiography is performed.

Exclusion Criteria:

Patients with:

* Life expectancy of less than one year.
* Previous AMI.
* Previous coronary revascularization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men and women undergoing coronary angioplasty.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2019-02-26 (Actual); Study Completion 2019-02-26 (Actual)

PRIMARY OUTCOMES:
Door-to-balloon time in patients | 90 minutes
  Door-to-balloon time in patients
Door-to-needle time in patients | 90 minutes
  Door-to-balloon time in patients
Time from onset of chest pain to first medical care | 24 hours
  Time from onset of chest pain to first medical care
Time from onset of chest pain to arrival Cath Lab | 24 hours
  Time from onset of chest pain to arrival Cath Lab
Time from onset of chest pain to artery opening | 24 hours
  Time from onset of chest pain to artery opening
Markers successful myocardial reperfusion by angiography | First 90 min after reperfusion.
  ST segment resolution 90 minutes post-PCI (Percutaneous Coronary Intervention)
Markers successful myocardial reperfusion by angiography | First 90 min after reperfusion.
  Final TIMI (Thrombolysis in Myocardial Infarction) flow grade
Markers successful myocardial reperfusion by angiography | First 90 min after reperfusion.
  Final TIMI blush grade
Underlying coronary anatomy assessment | 24 hours
  Final TIMI Thrombus grade
Underlying coronary anatomy assessment | 24 hours
  Degree of difuse disease
Underlying coronary anatomy assessment | 24 hours
  Number of vessels involve
Underlying coronary anatomy assessment | 24 hours
  Percentage of Ventricular Ejection Fraction
Underlying coronary anatomy assessment | 24 hours
  Presence of significant Left Main disease
Underlying coronary anatomy assessment | 24 hours
  Degree of distal embolization

SECONDARY OUTCOMES:
Major adverse cardiac events (MACE) | Hospital discharge and expected average of 1 week, one year follow-up
  MACE rate during hospitalization, defined as death, non-fatal myocardial rupture, or appearance or worsening of heart failure during the hospitalization period and after 1 year of follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitari Vall d'Hebron, Barcelona, Spain

REFERENCES:
- [Background] Writing Group Members; Mozaffarian D, Benjamin EJ, Go AS, Arnett DK, Blaha MJ, Cushman M, Das SR, de Ferranti S, Despres JP, Fullerton HJ, Howard VJ, Huffman MD, Isasi CR, Jimenez MC, Judd SE, Kissela BM, Lichtman JH, Lisabeth LD, Liu S, Mackey RH, Magid DJ, McGuire DK, Mohler ER 3rd, Moy CS, Muntner P, Mussolino ME, Nasir K, Neumar RW, Nichol G, Palaniappan L, Pandey DK, Reeves MJ, Rodriguez CJ, Rosamond W, Sorlie PD, Stein J, Towfighi A, Turan TN, Virani SS, Woo D, Yeh RW, Turner MB; American Heart Association Statistics Committee; Stroke Statistics Subcommittee. Executive Summary: Heart Disease and Stroke Statistics--2016 Update: A Report From the American Heart Association. Circulation. 2016 Jan 26;133(4):447-54. doi: 10.1161/CIR.0000000000000366. No abstract available. PMID 26811276
- [Background] 2. World Health Organization.The European Health Report2012: Chartingthe Wayto Well-being. Copenhagen, Denmark: World Health Organization Regional Office for Europe;2012
- [Background] Degano IR, Salomaa V, Veronesi G, Ferrieres J, Kirchberger I, Laks T, Havulinna AS, Ruidavets JB, Ferrario MM, Meisinger C, Elosua R, Marrugat J; Acute Myocardial Infarction Trends in Europe (AMITIE) Study Investigators. Twenty-five-year trends in myocardial infarction attack and mortality rates, and case-fatality, in six European populations. Heart. 2015 Sep;101(17):1413-21. doi: 10.1136/heartjnl-2014-307310. Epub 2015 Apr 8. PMID 25855798
- [Background] Garcia-Dorado D, Garcia del Blanco B. Door-to-balloon time and mortality. N Engl J Med. 2014 Jan 9;370(2):179. doi: 10.1056/NEJMc1313113. No abstract available. PMID 24401062
- [Background] Pancholy SB, Shantha GP, Patel T, Cheskin LJ. Sex differences in short-term and long-term all-cause mortality among patients with ST-segment elevation myocardial infarction treated by primary percutaneous intervention: a meta-analysis. JAMA Intern Med. 2014 Nov;174(11):1822-30. doi: 10.1001/jamainternmed.2014.4762. PMID 25265319